CLINICAL TRIAL: NCT05344001
Title: Life After Sport: Prior Injury and Sedentary Behavior as Mechanisms of Later Poor Health
Status: Recruiting | Type: Observational
Sponsor: Marquette University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 3967; DP5OD031833 (NIH)
Record Dates: First submitted 2022-04-12; First posted 2022-04-25 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Aging; Athletic Injuries; Physical Inactivity; Knee Injuries and Disorders
Keywords: Sports Medicine; Injury; Athlete; Sport; Physical Activity; Function; Health; Knee
MeSH Terms: conditions — Athletic Injuries; Sedentary Behavior; Knee Injuries; Disease; Wounds and Injuries; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Midlife former athletes with a prior knee injury: Inclusion Criteria: Age 40-64 years. Prior participation in a collision, contact, or jumping/cutting/pivoting sport (e.g., baseball, basketball, field hockey, football, ice hockey, lacrosse, soccer, softball, volleyball, etc.) at the collegiate varsity level for at least 1 season; history of at least 1 prior traumatic knee injury including but not limited to ACL or PCL rupture and/or reconstruction, medial and/or lateral meniscus tear or surgery, osteochondral defect, and/or intra-articular (i.e., tibiofemoral or patellofemoral) fracture.
  Exclusion Criteria: Neurologic (e.g., stroke, Parkinson's) and/or degenerative disease that impairs function; current pregnancy; lower extremity joint replacement (e.g., hip or knee replacement).
- Midlife former athletes without a prior major lower extremity injury: Inclusion Criteria: Age 40-64 years. Prior participation in a collision, contact, or jumping/cutting/pivoting sport (e.g., football, baseball, basketball, field hockey, ice hockey, lacrosse, soccer, softball, volleyball, etc.) at the collegiate varsity level for at least 1 season.
  Exclusion Criteria: Neurologic (e.g., stroke, Parkinson's) and/or degenerative disease that impairs function; current pregnancy; lower extremity joint replacement (e.g., hip or knee replacement); prior major lower extremity injury (e.g., ACL tear, Achilles tendon rupture, compound ankle or femur fracture, hip dislocation).
- Midlife controls: Inclusion Criteria: Age 40-64 years.
  Exclusion Criteria: Prior participation in a collegiate varsity sport or professional sport; neurologic (e.g., stroke, Parkinson's) and/or degenerative disease that impairs function; current pregnancy; lower extremity joint replacement (e.g., hip or knee replacement); prior major lower extremity injury (e.g., ACL tear, Achilles tendon rupture, compound ankle or femur fracture, hip dislocation).
- Young adult athletes: Inclusion Criteria: Age 18-25 years. Participation in a collision, contact, or jumping/cutting/pivoting sport (e.g., baseball, basketball, field hockey, football, ice hockey, lacrosse, soccer, softball, volleyball, etc.) at the varsity collegiate level.
  Exclusion Criteria: Neurologic (e.g., stroke, Parkinson's) and/or degenerative disease that impairs function; current pregnancy; lower extremity joint replacement (e.g., hip or knee replacement).
- Young adult controls: Inclusion Criteria: Age 18-25 years.
  Exclusion Criteria: Prior or current participation in any collegiate varsity sport; prior major lower extremity injury or surgery (e.g., ACL tear, Achilles tendon rupture, compound ankle or femur fracture, hip dislocation); current participation in competitive sport (e.g., collegiate club sport) more than 3x/week; joint replacement in the lower extremity (i.e., knee or hip replacement); current pregnancy; or neurologic condition (e.g., stroke, Parkinson's) and/or degenerative condition that impairs function.

SUMMARY:
Competitive sport increases risk for musculoskeletal injury (e.g., traumatic knee injury) and may position former athletes for early onset of chronic diseases, chronic pain, poor health-related quality of life, and disability. Quantifying function in former athletes with and without a prior injury and non-athlete controls is critical to understanding long-term health trajectories in athletes and informing potential interventional studies. One modifiable factor that may be associated with long-term health in athletes is physical activity patterns. The purpose of this study is to evaluate strength, function, physical activity, dietary patterns, and cardiometabolic health among current and former competitive athletes and in nonathlete controls to evaluate the impact of prior knee injury and sedentary behavior as two potential determinants of later poor health and reduced function.

DETAILED DESCRIPTION:
The overarching hypothesis is that former athletes, especially those with a prior injury, will have poorer function and health in midlife and that current and former athletes will engage in greater overall and longer bouts of sedentary behavior compared to non-athletes.

Aim 1 will compare function, strength, and cardiometabolic indicators among former athletes with and without prior knee injury and non-athlete controls in midlife (age 40-64). Hypothesis 1 is that former athletes with a prior injury will have the poorest function, muscle strength, and cardiometabolic indicators.

Aim 2 will compare sedentary behavior and physical activity patterns in current (age 18-25) and midlife former athletes to non-athlete controls. Hypothesis 2.1 is that current athletes will have greater sedentary behavior, longer sedentary behavior bouts, and higher levels of moderate-to-vigorous physical activity compared to non-athlete controls. Hypothesis 2.2 is that former athletes in midlife will have greater sedentary behavior, longer sedentary behavior bouts, and lower physical activity levels compared to non-athlete controls.

An exploratory aim will evaluate longitudinally the trajectory of physical activity patterns, cardiometabolic indicators, function, and strength annually in each cohort, comparing how these variables change over time in each subgroup.

ELIGIBILITY:
Please see cohorts for specific inclusion/exclusion criteria

Inclusion Criteria:

* Age 18-25 years OR age 40-64 years
* Current or former collegiate varsity athlete OR non-athlete control

Exclusion Criteria:

* Neurologic (e.g., stroke, Parkinson's) and/or degenerative disease that impairs function
* Pregnancy
* Lower extremity joint replacement (e.g., hip or knee replacement)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Current and former collegiate varsity athletes with and without a prior history of traumatic knee injury and matched non-athlete controls.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2022-04-18 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
30-Second Chair Stand Test (primary outcome for Aim 1) | Baseline
  Physical function (functional performance) will be evaluated using the 30-Second Chair Stand Test, 6-Minute Walk Test, and Stair Climb Test. The 30-Second Chair Stand Test uses a standard height chair and requires the participant to stand up and sit down as many times as possible in 30 seconds. More completions indicate better physical function.
Sedentary Behavior (primary outcome for Aim 2) | Baseline
  Physical activity will be monitored continuously using an accelerometer worn for 2 weeks. Physical activity will be classified throughout the day as sedentary, light, moderate, or vigorous using established algorithms. The primary outcome for aim 2 is the mean percentage of waking hours in sedentary behavior.

SECONDARY OUTCOMES:
Strength | Baseline
  Isometric quadriceps and hamstring strength will be assessed using a standardized strength testing machine (i.e., electromechanical dynamometer).
Body Composition | Baseline
  Body composition (i.e., percent body fat) will be assessed via dual-energy x-ray absorptiometry (DXA).
Step Counts | Baseline
  Average daily step counts will also be recorded using an objective physical activity monitor.
Cardiovascular Disease Risk | Baseline
  The American College of Cardiology/American Heart Association Atherosclerotic Cardiovascular Disease Risk Estimator will be used in the midlife participants to estimate 10-year cardiovascular disease risk.
6-Minute Walk Test | Baseline
  The 6-Minute Walk Test evaluates the distance participants can walk in 6 minutes and is a widely used indicator of function and aerobic capacity. The 6-minute walk test will be evaluated in the midlife participants only.
Stair Climb Test | Baseline
  The Stair Climb Test assesses the time it takes the participant to ascend and descend a flight of stairs. Faster times on the Stair Climb Test are associated with better strength and function. The Stair Climb Test will be evaluated in the midlife participants only.
Sedentary Behavior (follow-up) | Follow-up (an average of 1 year post-baseline)
  Physical activity will be monitored continuously using an accelerometer worn for 2 weeks. Physical activity will be classified throughout the day as sedentary, light, moderate, or vigorous using established algorithms. Mean percentage of waking hours in sedentary behavior and each physical activity classification will be assessed.
30-Second Chair Stand Test (follow-up) | Follow-up (an average of 1 year post-baseline)
  The 30-Second Chair Stand Test uses a standard height chair and requires the participant to stand up and sit down as many times as possible in 30 seconds. More completions indicate better physical function.
Strength (follow-up) | Follow-up (an average of 1 year post-baseline)
  Isometric quadriceps and hamstring strength will be assessed using a standardized strength testing machine (i.e., electromechanical dynamometer).
Body Composition (follow-up) | Follow-up (an average of 1 year post-baseline)
  Body composition (i.e., percent body fat) will be assessed via dual-energy x-ray absorptiometry (DXA).
Step Counts (Follow-up) | Follow-up (an average of 1 year post-baseline)
  Average daily step counts will also be recorded using an objective physical activity monitor.
6-Minute Walk Test (follow-up) | Follow-up (an average of 1 year post-baseline)
  The 6-Minute Walk Test evaluates the distance participants can walk in 6 minutes and is a widely used indicator of function and aerobic capacity. The 6-minute walk test will be evaluated in the midlife participants only.
Stair Climb Test (follow-up) | Follow-up (an average of 1 year post-baseline)
  The Stair Climb Test assesses the time it takes the participant to ascend and descend a flight of stairs. Faster times on the Stair Climb Test are associated with better strength and function. The Stair Climb Test will be evaluated in the midlife participants only.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob J. Capin, DPT, PhD, MS, Principal Investigator — Marquette University
Locations (1):
- Marquette University, Milwaukee, Wisconsin, United States

REFERENCES:
- See also: Official website of the Life After Sport Trajectories (LAST) Lab at Marquette University. — http://www.lastlab.org